CLINICAL TRIAL: NCT02339350
Title: Treatment of Newly Diagnosed High Risk Acute Lymphoblastic Leukemia in Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Korean Society of Pediatric Hematology Oncology (Network)
Responsible Party: Principal Investigator, Hee Young Shin, KSPHO, The Korean Society of Pediatric Hematology Oncology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSPHO_HRALL
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Acute Lymphoblastic Leukemia; Child
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rapid early responder group (No Intervention): 1. RER Consolidation BM exam on day 63: M1, M2 -> IM M3 or residual CNS ds or Bx proven extramedullary ds - off protocol
  2. RER Interim Maintenance #1
  3. RER Delayed Intensification
  4. RER Interim Maintenance #2
  5. RER Maintenance (12 weeks=84 days)
- Slow early responder group (Experimental): Includes : SER, Testis(+), CNS 3, T-cell (non ETP), Initial PB WBC ≥ 100,000/μL
  1. SER Consolidation
  * Intrathecal triple chemotherapy at d0, 7, 14, 21 2. SER Interim Maintenance #1
  * high dose methotrexate included
  * Intrathecal triple chemotherapy at d0, 28 3. SER Delayed Intensification #1
  * Intrathecal triple chemotherapy at d0, 28, 35 4. SER Interim Maintenance #2
  * high dose methotrexate included
  * Intrathecal triple chemotherapy at d0, 28 5. SER Delayed Intensification #2
  * Intrathecal triple chemotherapy at d0, 28, 35 6. SER Maintenance
  * Intrathecal triple chemotherapy at d0
  Interventions: Drug: high dose methotrexate; Drug: Intrathecal triple chemotherapy

INTERVENTIONS:
Drug: high dose methotrexate — HD-MTX IV 5,000 mg/m2 I.V. over 4hr on day 0, 14, 28, 42 of SER interim maintenance schedule
  Arms: Slow early responder group
Drug: Intrathecal triple chemotherapy — Intrathecal triple chemotherapy for SEG group instead of radiotherapy
  Arms: Slow early responder group

SUMMARY:
Treatment of pediatric acute lymphoblastic leukemia (ALL) has advanced and the overall survival exceeds 80% nowadays. However the overall survival of high risk ALL remains 75-90%, thus recent studies focus on treatment intensification according to the risk group. According to the previous reports, we designed a multicenter prospective trial for pediatric ALL.

DETAILED DESCRIPTION:
Purpose of the study

1. For slow early responder (SER), to confirm if the augmented interim maintenance using intravenous high dose methotrexate will improve the treatment outcome.
2. For slow early responder (SER), to confirm if removal of prophylactic radiotherapy will relieve long term complications.
3. To predict the treatment response and prognosis high risk pediatric ALL by monitoring of minimal residual disease (MRD).

Inclusion criteria

1. Diagnosis

1. Newly diagnosed B-precursor ALL meeting criteria 1.2
2. Newly diagnosed B-precursor ALL who was previously treated with steroid.
3. Newly diagnosed T cell ALL, excluding early T-cell precursor (ETP) leukemia

1.2 Initial WBC count

1. from 1 years old to 9 years old : WBC ≥ 50,000/μL
2. from 10 years old to 21 years old : Any WBC
3. from 1 years old to 21 years old : Any WBC with Testicular leukemia or CNS leukemia (CNS3)

Exclusion criteria (who are classified as very high risk group) 2.1 Philadelphia chromosome (+) or bcr/abl rearrangement (+) 2.2 Chromosome <45 by cytogenetics 2.3 Induction failure (Day 28 M3 marrow (>25% blasts)) 2.4 t(4:11) (as identified by cytogenetics, FISH or molecular studies) 2.5 Early T-cell precursor leukemia 2.6 Down syndrome ALL

Methods We will classify the patients to rapid early responder (RER) and slow early responder (SER), according to the treatment response after induction remission and risk factors at diagnosis. SER includes M2 (5-25% or leukemic cells at bone marrow exam) or M3 (25% or more of leukemic cells at bone marrow exam) response at the 14th day of the start of induction remission. If a patient showed total WBC count ≥ 100,000/μL, had testis or CNS (CNS 3) involvement at diagnosis and was diagnosed as T-ALL, the patients will also be included into the SER group.

Rapid early responders will undergo interim maintenance two times and reinduction for one time. Slow early responders will undergo two times of interim maintenance treatment with high dose intravenous methotrexate. For SER, adriamycin was previously administered only when absolute neutrophil count and platelet was normal, but it will be administered without restriction in this study. Both groups (RER and SER) will undergo maintenance chemotherapy thereafter, with the treatment duration of 3 years from the 1st interim maintenance for boys and 2 years for girls.

For SER group, prophylactic radiotherapy will not be done and it will be replaced by high dose intravenous methotrexate and intensification of intrathecal chemotherapy by replacing the intrathecal methotrexate to intrathecal cytarabine, methotrexate and hydrocortisone.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis

1. Newly diagnosed B-precursor ALL meeting criteria 1.2
2. Newly diagnosed B-precursor ALL who was previously treated with steroid.
3. Newly diagnosed T cell ALL, excluding early T-cell precursor (ETP) leukemia

1.2 Initial WBC count

1. from 1 years old to 9 years old : WBC ≥ 50,000/μL
2. from 10 years old to 21 years old : Any WBC
3. from 1 years old to 21 years old : Any WBC with Testicular leukemia or CNS leukemia (CNS3)

Exclusion Criteria:

1. Philadelphia chromosome (+) or bcr/abl rearrangement (+)
2. Chromosome <45 by cytogenetics
3. Induction failure (Day 28 M3 marrow (>25% blasts))
4. t(4:11) (as identified by cytogenetics, FISH or molecular studies)
5. Early T-cell precursor leukemia
6. Down syndrome ALL

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-01; Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
event-free survival of SER group | 5 years from diagnosis

SECONDARY OUTCOMES:
Number of adverse events | 5 years from diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University, College of Medicine, Seoul, South Korea